CLINICAL TRIAL: NCT02029326
Title: Biomarker Analysis in Metastatic Colorectal Cancer Treated With Cetuximab
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Joon Oh Park, MD, PhD, Samsung Medical Center
Other Study IDs: 2009-09-074
Record Dates: First submitted 2013-09-05; First posted 2014-01-07 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer, cetuximab, biomarker, prometheus
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Prometheus's Onco dX assay platform provides technological breakthrough for immunoassay by obtaining a level of sensitivity down to single tumor cells without compromising specificity. This allows assessment of multiple TKI treatment targets, their activation status, as well as down stream signaling proteins using very tiny amount of tissue that can be obtained by FNA or CTCs.

We planned this study to explore biomarkers predictive of clinical response to cetuximab-based treatment in metastatic colorectal cancer using the Prometheus Platform. We will also elucidate signal transduction pathway attributable to cetuximab resistance, monitor changes in the RTK activation status during cetuximab treatment using circulating tumor cells and analyze correlation between the quantity of circulating tumor cells and treatment response to cetuximab.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed metastatic colorectal cancer
* Cetuximab-based chemotherapy (monotherapy, combination therapy with cytotoxic chemotherapy such as FOLFOX, XELOX, irinotecan, FOLFIRI, XELIRI, first-line, second-line or third-line are all eligible)
* Age > 18 years.
* ECOG Performance Status of 0-2
* Adequate bone marrow, liver and renal function
* Signed and dated informed consent before the start of specific protocol procedures.
* FNA will be performed in patients with feasible biopsy site; ascites or pleural fluid will be collected in metastatic CRC patients with ascites or pleural effusion

Exclusion Criteria:

* Active clinically serious infections (> grade 2 CTCAE version 3.0)
* Patients with evidence or history of bleeding diathesis
* Radiotherapy during study or within 4 weeks of start of study drug.
* Prior exposure to the study drug.
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: colorectal cancer patients who are treated with cetuximab
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-08-26 (Actual)

PRIMARY OUTCOMES:
To explore biomarkers predictive of clinical response to cetuximab-based treatment in metastatic colorectal cancer using the Prometheus Platform | at Screening (Day - 21 ~ 0 ), at 4 weeks and average 6months(end of treatment)
  A. To analyze expression and activation status of receptor tyrosine kinases in signal transduction pathways in FNA samples and circulating tumor cells B. To identify negative predictive markers to cetuximab

SECONDARY OUTCOMES:
1. RTK activation status during cetuximab treatment using circulating tumor cells | at Screening (Day - 21 ~ 0 ), at 4 weeks and average 6months(end of treatment)
2. signal transduction pathway attributable to cetuximab resistance | at Screening (Day - 21 ~ 0 ), at 4 weeks and EOT (end of treatment)
3. To analyze correlation between the quantity of circulating tumor cells and treatment response to cetuximab | at Screening (Day - 21 ~ 0 ), at 4 weeks and average 6months (end of treatment)

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea